CLINICAL TRIAL: NCT04524702
Title: Phase II Trial of Paricalcitol and Hydroxychloroquine (PH) Combination With Gemcitabine and Nab-Paclitaxel in Advanced or Metastatic Pancreatic Cancer
Brief Title: Paricalcitol and Hydroxychloroquine in Combination With Gemcitabine and Nab-Paclitaxel for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000996; NCI-2020-05417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship5079-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-08-13; First posted 2020-08-24 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Advanced Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Hydroxychloroquine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paricalcitol, hydroxychloroquine, chemotherapy) (Experimental): Beginning day -14, patients receive paricalcitol IV three times weekly and hydroxychloroquine PO BID. Patients also receive gemcitabine IV over 30 minutes and nab-paclitaxel IV over 30 minutes on days 1, 8, 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Hydroxychloroquine; Drug: Nab-paclitaxel; Drug: Paricalcitol

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Hydroxychloroquine — Given PO
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Drug: Paricalcitol — Given IV
  Other Names: Compound 49510; Zemplar

SUMMARY:
This phase II trial investigates how well paricalcitol and hydroxychloroquine work when combined with gemcitabine and nab-paclitaxel in treating patients with pancreatic cancer that has spread to other places in the body (advanced or metastatic). Paricalcitol (a form of vitamin D) works by blocking a signal in the cancer cells that leads to growth and spreading of the tumor. Hydroxychloroquine (an autophagy inhibitor) enhances the activity of standard chemotherapy on cancer cells and prevent them to utilize energy to grow. Chemotherapy drugs, such as gemcitabine and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving paricalcitol and hydroxychloroquine together with standard chemotherapy (gemcitabine and nab-paclitaxel) may work better in treating patients with pancreatic cancer compared to either paricalcitol or hydroxychloroquine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the anti-tumor activity of the combination of paricalcitol plus hydroxychloroquine (PH) when added to gemcitabine and nab-paclitaxel treatment by assessing the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of paricalcitol plus hydroxychloroquine (PH) when added to gemcitabine and nab-paclitaxel treatment in patients with advanced pancreatic cancer.

II. To evaluate the anti-tumor activity of the combination of paricalcitol plus hydroxychloroquine (PH) when added to gemcitabine and nab-paclitaxel treatment by assessing progression-free survival (PFS) and overall survival (OS).

TERTIARY/EXPLORATORY OBJECTIVES:

I. Evaluate the effects of PH on cancer-associated fibroblasts (CAF) and immune cells using mass cytometry (CyTOF) to characterize the presence and distribution of these cells.

II. Multiplex immunohistochemistry (IHC) to evaluate these pathways including TGF-beta1, TGF-beta1 RII, SMAD4, LC3 in addition to markers of fibrosis (collagen) and tumor (cytokeratin).

OUTLINE:

Beginning day -14, patients receive paricalcitol intravenously (IV) three times weekly and hydroxychloroquine orally (PO) twice daily (BID). Patients also receive gemcitabine IV over 30 minutes and nab-paclitaxel IV over 30 minutes on days 1, 8, 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced or metastatic adenocarcinoma of the pancreas (stage IV)
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded as >= 10 mm (>= 1 cm) on computed tomography (CT) scan, magnetic resonance imaging (MRI)
* Patients may have had prior neoadjuvant or adjuvant treatment for pancreatic cancer. The last dose of chemotherapy must have been 12 months prior to study entry. No prior systemic therapy for metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9.0 g/dl (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 28 days of cycle 1 day 1)
* Absolute neutrophil count (ANC) >= 1,500/mcL (after at least 7 days without growth factor support or transfusion) (within 28 days of cycle 1 day 1)
* Platelets >= 100,000/mcL (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 28 days of cycle 1 day 1)
* International normalized ratio (INR) =< 1.5 (within 28 days of cycle 1 day 1)
* Partial thromboplastin time (PTT) < 1.5 x upper limits of normal (ULN) (within 28 days of cycle 1 day 1)
* Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5.0 times the ULN (within 28 days of cycle 1 day 1)
* Serum creatinine =< 1.5× ULN or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x ULN. Creatinine clearance should be calculated per institutional standard (within 28 days of cycle 1 day 1)
* Calcium (corrected for albumin) =< 1 x institutional upper limit of normal (within 28 days of cycle 1 day 1)
* Patients with prior radiotherapy are acceptable. It must be at least 21 days since administration of radiation therapy and all signs of toxicity must have abated
* Patient must have a primary or metastatic non-bone site that is amenable to safe biopsy. Bone only lesions are not suitable for biopsy
* Patients with known G6PD deficiency, severe psoriasis, porphyria, macular degeneration or severe diabetic retinopathy are ineligible because of the potential for greater hydroxychloroquine (HCQ) toxicity
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardio- toxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of study drugs used in this study on the developing human fetus are unknown. For this reason, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 1 month after completion of drug administration
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Prior chemotherapy or any other investigational agents for the treatment of metastatic pancreatic cancer
* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents
* History of use of HCQ (aminoquinolines) or paricalcitol in the 6 months prior to study entry
* Pre-existing hypercalcemia, defined as baseline serum calcium (corrected for albumin) above the institutional upper limit of normal
* After signing consent, vitamin D or calcium containing supplements must be stopped and no vitamin D or calcium supplements can be taken while the patient is enrolled to the study due to increased risk for hypercalcemia
* Pre-existing, clinically significant peripheral neuropathy, defined as Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher neurosensory or neuro-motor toxicity, regardless of etiology
* Participants with uncontrolled brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Current use of medications that prolong QT interval unless approved by principal investigator (PI) or substances that are strong inhibitors or inducers of CYP450 3A enzyme(s)- unless approved by PI
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with known G6PD deficiency, severe psoriasis, porphyria, macular degeneration or severe diabetic retinopathy are ineligible because of the potential for greater HCQ toxicity
* Pregnant women are excluded from this study because the use of agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs, breastfeeding should be discontinued
* Participant must be able to swallow and absorb pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji B. Alese, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hosptial, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagaraju GP, Saddala MS, Foote JB, Khaliq AM, Masood A, Golivi Y, Bandi DSR, Sarvesh S, Reddy SP, Switchenko J, Carstens JL, Akce M, Herting C, Alese OB, Yoon KJ, Manne U, Bhasin MK, Lesinski GB, Sukhatme VP, El-Rayes BF. Mechanism of enhancing chemotherapy efficacy in pancreatic ductal adenocarcinoma with paricalcitol and hydroxychloroquine. Cell Rep Med. 2025 Jan 21;6(1):101881. doi: 10.1016/j.xcrm.2024.101881. Epub 2024 Dec 26. PMID 39730001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Tumor Response to Combination of Paricalcitol and Hydroxychloroquine With Common Front-line Therapy.
Description: To evaluate the anti-tumor activity of the combination of paricalcitol plus hydroxychloroquine (PH) when added to gemcitabine and nab-paclitaxel treatment by assessing the Overall Response Rate (ORR) by RECIST 1.1. ORR is defined as the percentage of people in the trial who have partial response (PR) or complete response (CR). The Response rate will be estimated with Clopper-Pearson with a 90% exact confidence interval.
Time Frame: At 8 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 7
percentage of participants | 43 [10 to 82]

2. Secondary Outcome: Incidence of Adverse Events
Description: Toxicities will be presented as worst toxicity per patient and will be reported as percent toxicity. The number of subjects with skipped doses, dose delays and dose reductions as well as major reasons for dose modifications will be summarized. Adverse events will be classified using MedDRA System Organ Classes and Preferred Terms. Furthermore, serious adverse events (SAEs), adverse events (AEs) with a severity grade of 3 or above using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, AEs deemed related to study drug, AEs leading to discontinuation of study drug, and AEs leading to death will also be summarized in preferred term by system organ class and listed on an individual subject basis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 9
Participants
  Action taken after AE, No action taken | 7
  Action taken after AE, dose interrupted | 2
  Action taken after AE, dose decreased | 0
  Action taken after AE, discontinued | 0

3. Secondary Outcome: Progression-free Survival
Description: Assessed using RECIST 1.1. Will be estimated using the Kaplan-Meier method.
Time Frame: 32.5 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 10
months | 6 [1.4 to 6.7]

4. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: 32.5 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 7
Months | 6.8 [1.8 to 9.9]

5. Other Pre Specified Outcome: Percentage Change in Circulating Pancreatic Ductal Adenocarcinoma Cells
Description: Will evaluate changes in immune and malignant circulating cells before and after treatment with PH when added to gemcitabine and nab-paclitaxel treatment and their relationship.
Time Frame: blood collection was done at baseline (day -7), cycle 2 day 1.
Measure: Mean (Standard Deviation); unit: percentage change in PDAC cells
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
Number analyzed (Participants) | 7
percentage change in PDAC cells | 50 (0.5)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy) (N=10)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paricalcitol, Hydroxychloroquine, Chemotherapy) (N=10)
Nausea (Gastrointestinal disorders) | 7 (14)
anemia (Blood and lymphatic system disorders) | 7 (40)
Thromboembolic Event (Blood and lymphatic system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 9 (13)
Fatigue (General disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (5)
Hypercalcemia (Investigations) | 3 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Neutropenia (Investigations) | 3 (3)
Leukopenia (Investigations) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04524702/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04524702/ICF_001.pdf